CLINICAL TRIAL: NCT00402454
Title: Evaluation of Three Regimens of Chemoprophylaxis for Tuberculosis in Patients co-Infected by HIV and Mycobacterium Tuberculosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAEI 94/0071B; FIS 94/0071B
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections
Keywords: HIV; Tuberculosis; Prophylaxis; AIDS
MeSH Terms: conditions — HIV Infections; Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — Isoniazid; Rifampin; Pyrazinamide

INTERVENTIONS:
Drug: isoniazid, rifampin + isoniazid or rifampin + pyrazinamide

SUMMARY:
To evaluate adherence and safety of three regimens of chemoprophylaxis for tuberculosis (TB) in HIV-infected patients with positive tuberculin skin test.

DETAILED DESCRIPTION:
DESINGS: We performed a randomised, comparative and open clinical assay carried out in 316 HIV-infected patients. The patients were randomly assigned to one of three regimens, 108 to isoniazid for six months (6H), 103 to rifampin and isoniazid for three months (3RH), and 105 to pyrazinamide and rifampin for two months (2RZ).

RESULTS: The TB rates (cases per 100 persons/year) in the three treatment groups were 3.4 in 6H, 4.5 in 3RH and 1.9 in 2RZ. The relative risk for TB with 6H as compared with 2RZ was 1.76, and with 3RH, 2.34. Twenty-seven percent of the patients voluntarily abandoned chemoprophylaxis and 9.7% were withdrawn due to adverse side-effects. Seven patients were withdraw due to hepatotoxicity (5 in 6H, 2 in 3RH and 0 in 2RZ). No appreciable differences were found among the three regimens.

CONCLUSION: In our study the 2RZ regimen was as safe as the 6H and 3RH regimens. We have nor observed a higher incidence of hepatotoxicity in patients who received 2RZ.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection confirmed by ELISA and Western blot
* Age between 18 and 65 years
* Life expectancy greater than two years
* Reactivity to PPD > 5 mm

Exclusion Criteria:

* Presence of active tuberculosis
* Background of previous antituberculosis therapy or chemoprophylaxis
* Presence of symptoms or signs suggesting pulmonary or extra-pulmonary tuberculosis
* History of hypersensitivity to the drugs used in the study (isoniazid, rifampin or pyrazinamide)
* Aspartate-aminotransferase and/or alanine-aminotransferase plasma concentrations more than or equal to four times their normal values, total bilirubin more than 2 mg/ml, and/or creatinine more than 2 mg/ml
* Pregnancy
* Undergoing treatment incompatible with any of the drugs used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1994-01; Study Completion 1998-12

PRIMARY OUTCOMES:
Development of Tuberculosis
Suspension of chemoprophylaxis due to adverse effects

SECONDARY OUTCOMES:
Suspension of chemoprophylaxis due tovoluntary withdrawal
Mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rivero, MD PhD, Study Chair — Hospital Universitario Reina Sofía, Córdoba, Spain; Luis Lopez-Crtés, MD, PhD, Principal Investigator — Hospital Universitario Virgen del Rocío, Sevilla, Spain; Rafael Castillo, MD, Principal Investigator — 3 Sección de Enfermedades Infecciosas. Hospital Clínico Universitario San Cecilio. Avda. Dr. Oloriz 16. 18012 Granada; José Verdejo, MD, Principal Investigator — Servicio de Enfermedades Infecciosas. Hospital Carlos III. Sinesio Delgado 10. 28029 Madrid; Miguel Angel García, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Carlos Haya. Avda. Carlos Haya s/n. 29010 Málaga.; Felipes Diez, MD, Principal Investigator — Servicio de Medicina Interna. Hospital Torrecárdenas. Paraje de Torrecárdenas s/n. 04009 Almería.; Jose Carlos Escribano, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Puerta del Mar. Avda. Ana de Viya, 21. 11009 Cádiz. Spain; Jesús Canueto, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Punta Europa de Algeciras. Ctra de Getares s/n. 11207 Algeciras (Cádiz)., Spain; Manuel Marquez, MD, Principal Investigator — Unidad de Enfermedades Infecciosas. Hospital Universitario Virgen de la Victoria, Campus Universitario Teatinos s/n. 29010 Málaga.; Juan Jose Hernandez, MD, Principal Investigator — Unidad de Enfermedades Infecciosas. Hospital Ciudad de Jaén, Avda del Ejército Español, 10. 23007 Jaén, Spain.; Juan Pasquau, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Virgen de las Nieves. Avda de las Fuerzas Armadas, 2. 18014 Granada, Spain.; Fernando Lozano, MD PhD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Virgen de Valme. Ctra. de Cádiz s/n. 41012 Sevilla, Spain
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain